CLINICAL TRIAL: NCT01737749
Title: Validation of Neurokeeper's Algorithm on Patients Undergoing Cardiac Surgery.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neurokeeper Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: NK-005
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgery
  Interventions: Device: Neurokeeper stroke detector

INTERVENTIONS:
Device: Neurokeeper stroke detector — Electrophisoloigcal monitoring

SUMMARY:
The primary objective of the study is to check the ability of Neurokeeper's algorithm system to detect and monitor changes in cerebral electrophysiological parameters as compared to clinical evaluation in patients undergoing cardiac surgery.

The secondary objectives is correlations of EEG + ERP measurements with clinical evaluations as assessed by NIHSS ThiS study is a prospective, open label, single arm, self control, single center study.

This study will be conducted in 50 subjects according to the inclusions/exclusions criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Patients undergoing cardiac surgery .

Exclusion Criteria:

* Previous major hemispheric stroke.
* Any known major hemispheric lesion.
* Significant movement disorder.
* Local skull or skin affliction which prevents electrodes application.
* Any known condition which in the opinion of the investigator may interfere with the protocol implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Neurological detrioration detection
  The primary objective of the study is to validate an EEG base algorithm system to detect and monitor changes in cerebral electrophysiological parameters as compared to clinical evaluation in patients undergoing cardiac surgery.

SECONDARY OUTCOMES:
Time from deterioration to detection
  The secondary objectives is correlations of EEG + ERP measurements with clinical evaluations as assessed by NIHSS

CONTACTS AND LOCATIONS:
Overall Officials: Moshe' Herskovitz, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel